CLINICAL TRIAL: NCT01077869
Title: A Feasibility Study on the Use of F-18-FDG-PET and Optical Imaging in Evaluation of Radiation-induced Oral Mucositis
Status: Terminated | Type: Observational
Why Stopped: poor recruitment rate
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Wilfried De Neve, MD, PhD, University Hospital Ghent
Other Study IDs: 2009/621
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity; Oropharynx Metastases; Lymph Metastases
Keywords: oropharynx and lymph node metastases from an unknown primary tumor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: endoscopic examination — on a weekly basis during 7 weeks
Procedure: FDG-PET — once pre-radiotherapy and once 2 weeks after initiation of radiotherapy

SUMMARY:
In this study, the feasibility of optical imaging and FDG-PET in the evaluation of radiation-induced mucositis will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Non-operated histologically confirmed squamous cell carcinoma of the oral cavity, oropharynx (except the posterior wall) and lymph node metastases from the unknown primary tumor (CUP)
* Stage T1-4; Tx N+ for the CUP
* Multidisciplinary Group of Head and Neck Tumors at Ghent University Hospital decision of radical radiotherapy (±concurrent chemotherapy)
* Informed consent obtained, signed and dated before specific protocol procedures.

Exclusion Criteria:

* Age < 18 years
* Pregnant or lactating women
* Active infection or fistula in the oral/oropharyngeal mucosa
* Previous cancer of the oral cavity and the oropharynx
* Prior head-and-neck radiotherapy
* Expectation of non-compliance with the study protocol
* Known allergy for topical anesthetics (Xylocaïne)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Squamous cell carcinoma of the oral cavity, oropharynx and lymph node metastases from unknown primary tumor.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of optical imaging in the evaluation of radiation-induced mucositis. | weekly assessment during 7 weeks
Feasibility of FDG-PET in the evaluation of radiation-induced mucositis. | 2 weeks after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: wilfried De Neve, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be